CLINICAL TRIAL: NCT03315507
Title: An Open-Label, Dose Titration Study to Assess the Safety, Tolerability, and Hemodynamic Response of PB1046, A Sustained-Release Analogue of Vasoactive Intestinal Peptide, In Adult Subjects With Pulmonary Arterial Hypertension
Brief Title: A Study to Assess the Safety, Tolerability, and Hemodynamic Response of PB1046 in Subjects With PAH
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PhaseBio Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PB1046-PT-CL-0005
Record Dates: First submitted 2017-10-02; First posted 2017-10-20 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Intervention Model Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PB1046 Injection (Experimental): PB1046 Subcutaneous Injection
  Interventions: Drug: PB1046 Subcutaneous Injection

INTERVENTIONS:
Drug: PB1046 Subcutaneous Injection — Eight weekly doses of PB1046.

SUMMARY:
PB1046-PT-CL-0005 is an open-label, dose-titration study to assess the safety, tolerability, and hemodynamic effects of individually dose-titrated PB1046 administered by weekly subcutaneous injection for 8 weeks in adult subjects with PAH who have a permanently implanted hemodynamic monitor in the distal pulmonary artery. The primary objectives of the study are to assess the overall safety, tolerability, and hemodynamic profile of a PB1046 across an individually titrated dose range.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent and follow all study-related procedures;
* Confirmed diagnosis of Pulmonary Arterial Hypertension (WHO Group 1) and WHO Functional Class II or III by clinical diagnostic criteria assessed by the Investigator and have a permanently implanted pulmonary artery hemodynamic monitor (IHM);
* Adult subjects ≥18 years of age willing and able to utilize contraception as needed for 30 days after their last dose of study drug;
* Body mass index ≥ 18 kg/m2 and ≤ 47 kg/m2;
* Receipt of Investigator-directed stable (no change in dose or addition or removal of a therapy) medical-therapy in accordance with local standard of care for the management of PAH for 30 days prior to screening and between screening and first dose and are in stable clinical condition;
* Screening hemoglobin ≥ 9.0 g/dL secondary to the volume of blood to be collected during the study period;
* Willing and able to return to the study unit for specified study visits, or accommodate home visits;
* Willing and able to transmit hemodynamics via IHM and monitor systemic blood pressure while at home and record results.

Exclusion Criteria:

* Concomitant medical disorder, condition, or history, that in the opinion of the Investigator would impair the subject's ability to participate in or complete the requirements of the study;
* Concomitant medical disorder that is expected to limit the subject's life-expectancy to ≤ 1 year;
* Pregnant or lactating female subjects;
* First positive result from serology testing at visit 1 (screening labs) for human immunodeficiency virus, hepatitis B surface antigen, or hepatitis C virus prior to first dose;
* Participation in another investigational study within 30 days prior to screening or are taking part in a non-medication study which, in the opinion of the Investigator, would interfere with the study compliance or outcome assessments;
* Use of bosentan therapy for PAH within 30 days prior to screening or during study participation;
* Sustained systolic blood pressure (SBP) < 95 mmHg and/or diastolic blood pressure (DBP) < 50 mmHg (confirmed by a duplicate seated reading) on at least 3 consecutive readings (self-monitored or office) prior to first dose, or overt symptomatic hypotension;
* Sustained resting heart rate >110 beats per minute (BPM) at screening (V1) or prior to first dose (confirmed by duplicate assessments of office vital signs or consecutive ECG assessments) on at least 3 consecutive readings prior to first dose;
* Clinically significant renal dysfunction as measured by the estimated glomerular filtration rate (eGFR) of < 40 mL/min/1.73m2 as calculated by the MDRD equation: eGFR = 175 x (Creat / 88.4)-1.154 x (Age)-0.203 x (0.742 if female) x (1.212 if African American) (conventional units);
* Clinically significant liver dysfunction as measured by any one of the following: a. alanine aminotransferase (ALT) >3.0 time ULN or; b. aspartate aminotransferase (AST) >3.0 time ULN or; c. serum bilirubin ≥ 1.6 mg/dL;
* Known history of substance abuse that in the opinion of the Investigator would impair the subject's ability to participate in or complete the requirements of the study;
* Any major surgical procedure within 30 days prior to screening or planned surgical procedure during the study period;
* In-patient hospitalization (defined as greater than 23 hours) within 30 days of subject dosing;
* Enrollment within the past 3 months prior to screening or plans to enroll during the study into a cardiopulmonary rehabilitation program;
* Other medical or psychiatric condition which, in the opinion of the Investigator, would place the subject at increased risk or would preclude obtaining voluntary consent or would confound the objectives of study;
* Known hypersensitivity to study drug or any of the excipients of the drug formulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2019-08-08 (Actual); Study Completion 2019-08-08 (Actual)

PRIMARY OUTCOMES:
Adverse Events | Pre-dose to 28 days after last dose
  Incidence and severity of AEs (described descriptively) and their relationship to study drug
Vital Signs (Blood pressure) | Prior to eight weekly doses and 1 and 3 hours after the final dose and 1, 2, 3, 5, 7 and 28 days after final dose.
  Changes from baseline in blood pressure and their relationship to study drug
Vital Signs (Heart rate) | Prior to eight weekly doses and 1 and 3 hours after the final dose and 1, 2, 3, 5, 7 and 28 days after final dose.
  Changes from baseline in heart rate and their relationship to study drug
Laboratory Parameters (Lipids) | Pre-dose and 7 and 28 days after last dose
  Changes from baseline in lipids and their relationship to study drug
Laboratory Parameters (Serum chemistry) | Pre-dose and prior to doses 2-8 and 7 and 28 days after last dose
  Changes from baseline in serum chemistry and their relationship to study drug
Laboratory Parameters (Urinalysis) | Pre-dose and prior to doses 2-8 and 7 and 28 days after last dose
  Changes from baseline in urinalysis and their relationship to study drug
Laboratory Parameters (NT-pro-BNP) | Prior to doses 1-8 and 7 and 28 days after last dose
  Changes from baseline in NT-pro-BNP and their relationship to study drug
Mean Pulmonary Artery Pressure | Prior to eight weekly doses and 1 and 3 hours after the final dose and 1, 2, 3, 5, 7, 8 and 28 days after final dose
  Change from baseline in mean pulmonary artery pressure
Cardiac Index | Prior to eight weekly doses and 1 and 3 hours after the final dose and 1, 2, 3, 5, 7, 8 and 28 days after final dose
  Change from baseline in cardiac index
Total pulmonary resistance | Prior to eight weekly doses and 1 and 3 hours after the final dose and 1, 2, 3, 5, 7, 8 and 28 days after final dose
  Change from baseline in total pulmonary resistance
Laboratory Parameters (Fasting Plasma Glucose) | Pre-dose and 7 and 28 days after last dose
  Changes from baseline in fasting plasma glucose and their relationship to study drug
Laboratory Parameters (Hematology) | Pre-dose and prior to doses 2-8 and 7 and 28 days after last dose
  Changes from baseline in hematology and their relationship to study drug

SECONDARY OUTCOMES:
Pharmacokinetic Dose Exposures (AUC (0-t)) | Prior to eight weekly doses and at 1, 3, 24, 48, 72,120, 168 and 192 hours after final dose.
  Area under the curve over the dosing interval (AUC(0-t))
Pharmacokinetic Dose Exposures (AUC (0-tmax)) | Prior to eight weekly doses and at 1, 3, 24, 48, 72,120, 168 and 192 hours after final dose.
  Area under the curve concentration-time profile (AUC(0-tmax))
Pharmacokinetic Dose Exposures (Cmax) | Prior to eight weekly doses and at 1, 3, 24, 48, 72,120, 168 and 192 hours after final dose.
  Maximum serum concentration (Cmax)
Pharmacokinetic Dose Exposures (Tmax) | Prior to eight weekly doses and at 1, 3, 24, 48, 72,120, 168 and 192 hours after final dose.
  Time to Cmax (Tmax)
Pharmacokinetic Dose Exposures (Ctrough) | Prior to eight weekly doses and at 1, 3, 24, 48, 72,120, 168 and 192 hours after final dose.
  Pre-dose serum concentrations at Weeks 1 through 7 and the concentrations after the last dose
Pharmacokinetic Dose Exposures (t1/2) | Prior to eight weekly doses and at 1, 3, 24, 48, 72,120, 168 and 192 hours after final dose.
  Half-life (t1/2)
Pharmacokinetic Dose Exposures (Lambda z) | Prior to eight weekly doses and at 1, 3, 24, 48, 72,120, 168 and 192 hours after final dose.
  Lambda z
Pharmacokinetic Dose Exposures (Cl/F) | Prior to eight weekly doses and at 1, 3, 24, 48, 72,120, 168 and 192 hours after final dose.
  Apparent clearance (Cl/F)
Pharmacokinetic Dose Exposures (Vd/F) | Prior to eight weekly doses and at 1, 3, 24, 48, 72,120, 168 and 192 hours after final dose.
  Volume of distribution (Vd/F)
Immunogenicity | Prior to eight weekly doses and on study days 59, 77 and 105.
  Incidence of immunogenicity

OTHER OUTCOMES:
6 Minute Walk Distance Test (6MWD) | Pre-dose and 7 days after final dose
  Change from baseline in 6MWD
Borg Dyspnea Index (BDI) | Pre-dose and 7 days after final dose
  Change from baseline in BDI
PAH Related Biomarkers | Prior to Dose 1, prior to Dose 5 and 7 days after final dose
  Change from baseline in PAH related biomarkers

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Allegheny General Hospital, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No